CLINICAL TRIAL: NCT00533312
Title: A Multicenter, Randomized, Double-Blinded, Parallel-Design Study to Evaluate the Lipid-Altering Efficacy of 2 Formulations of MK0524A Compared to NIASPAN (TM)
Brief Title: MK0524A Clinical Efficacy Study (0524A-026)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0524A-026; 2007_619
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Niacin; MK-0524; Duration of Therapy

INTERVENTIONS:
Drug: Comparator : placebo (unspecified) / Duraton of Treatment: 4 Weeks
Drug: MK0524A, niacin (+) laropiprant / Duration of Treatment : 4 Weeks
Drug: Comparator : niacin / Duraton of Treatment: 4 Weeks

SUMMARY:
A study to determine lipid changing effects of MK0524A when compared to niacin extended release (NIASPAN) and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 and 70 years
* Female patients must be pre-menopausal women that have been surgically sterilized, not pregnant and/or not planning to become pregnant

Exclusion Criteria:

* Patient has a history of peptic ulcer or gout
* Patient is sensitive to niacin or products containing niacin
* Patient drinks more than 2 alcoholic drinks per day
* Patient has certain heart disease, cancer, or is HIV positive

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2005-04; Primary Completion 2005-07 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To assess the HDL-C raising efficacy of MK-0524A when compared with niacin extended release (NIASPAN) and placebo. | After 4 weeks

SECONDARY OUTCOMES:
To asses the triglyceride-lowering effects of MK-0524A when compared with niacin extended release (NIASPAN) and placebo. | After 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Lai E, De Lepeleire I, Crumley TM, Liu F, Wenning LA, Michiels N, Vets E, O'Neill G, Wagner JA, Gottesdiener K. Suppression of niacin-induced vasodilation with an antagonist to prostaglandin D2 receptor subtype 1. Clin Pharmacol Ther. 2007 Jun;81(6):849-57. doi: 10.1038/sj.clpt.6100180. Epub 2007 Mar 28. PMID 17392721
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html